CLINICAL TRIAL: NCT01750047
Title: A Epidemiological Survey of Preoperative Pain Perception and Postoperative Pain in Chinese Population
Status: Completed | Type: Observational
Sponsor: Xianwei Zhang (Other)
Responsible Party: Sponsor-Investigator, Xianwei Zhang, Clinical Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: Pain Epidemiology
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Pain; Surgery
Keywords: pain perception; postoperative pain; demography; smoking; alcohol
MeSH Terms: conditions — Pain; Pain, Postoperative; Smoking

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Object: Every person's pain perception and possible postoperative pain is different. As the investigators know, they are affected by many factors. However, the investigators don't know whether the smoking factors, alcohol factors, surgery type, education background, etc. will affect individual pain perception and possible postoperative pain in Chinese population. This study was conducted to investigate the power of these possible affect factors. Method: Patients receiving elective surgery under general anesthesia were recruited into this study. The investigators measured their preoperative pressure pain threshold (PPT) and pressure pain tolerance (PTO)and also investigated the patient's personal information of smoking factors, alcohol factors, surgery type, education background, etc. In addition, we retrospectively investigated the visual analog scale (VAS) during patient-controlled analgesia (PCA) treatment 0 to 48 h after operation as well as the PCA press frequency and drug consumption of those patients who received PCA administration.

DETAILED DESCRIPTION:
Patients with the following diseases were excluded: known history of chronic pain, psychiatric diseases or communication disorders, diabetes mellitus, severe cardiovascular diseases, kidney or liver diseases with poor hepatic function, alcohol or pregnancy or at the lactation period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70
* The right hand is handedness
* Agreed to participate the research
* Not with known chronic disease
* Not taking analgesics within 3 months

Exclusion Criteria:

* History of chronic pain diseases
* Diabetes mellitus
* Severe cardiovascular diseases
* Kidney or liver diseases
* Alcohol or drug abuse
* Pregnancy or at lactation period
* Disagree to participate to the research

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients receiving elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 1327 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | 1 year
Pressure pain tolerance | 1 year

SECONDARY OUTCOMES:
Pain scores on visual analog scale after operation | 1 year
Opioid consumption dose after operation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xianwei, Doctor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China